CLINICAL TRIAL: NCT01507155
Title: An Open Label Study of Clinical Utility and Patient Outcomes of the Genecept Assay
Acronym: COM-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genomind, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COM-1
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Treatment Resistant Depression; Generalized Anxiety Disorder
Keywords: Major; Depressive; Disorder; Depression; MDD; Treatment Resistant; Anxiety; GAD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Generalized Anxiety Disorder; Disease; Depression; Anxiety Disorders | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient-Reported Measures (Experimental): Patients age 18 and older with a diagnosis of Major Depressive Disorder or Generalized Anxiety disorder who received genetic testing using the Genecept Assay and completed patient scales.
  Interventions: Device: Genecept Assay
- Clinician-Reported Outcomes (Experimental): Prescribing clinicians responsible for the treatment of patients age 18 and older with a primary diagnosis of Major Depressive Disorder or Generalized Anxiety disorder, and for whom the Genecept Assay has been utilized to perform genetic testing.
  Interventions: Device: Genecept Assay

INTERVENTIONS:
Device: Genecept Assay — Genetic test which analyzes seven pharmacodynamic and three pharmacokinetic genes important in psychiatric disorders
  Other Names: Genetic Test

SUMMARY:
Genomind has developed and introduced a battery of genetic tests, the Genecept Assay, which clinicians can administer to patients using a simple saliva sample technique. The present study proposes to enroll 1. Subjects (patients who have consented to using the Genecept Assay) and 2. Clinician study participants (clinicians who have ordered the Assay on behalf of their patients). This study will involve the collection of responses from both Subjects and clinician study participants with the intention of correlating this information to Subject genetic data.

DETAILED DESCRIPTION:
This will be a 3-month prospective study of clinicians who have ordered the Genecept assay and the psychiatric patients for whom the test was ordered. Clinicians who order the Assay for a patient who has been indicated as having a diagnosis of depression will receive an invitation to participate in this study as well as an informational patient study brochure with the test kit. The patient's treating clinician will be prompted to discuss the study with the patient. Clinicians and patients can view a website containing additional information about the study as well as the informed consent document.

Potential subjects and clinician study participants will be consented online using a secure electronic method. Study staff will be available by phone and by email to answer any questions related to the study and the informed consent documents and process. Clinicians and patients can choose to participate independently of each other so that if one party declines to enroll, the other may still participate. Whether or not they choose to participate, patients must consent to allow their clinicians to provide responses about their treatment.

All subjects and participants will receive a username and password with which to access the secure study portal for completion of study surveys. Subjects and participants will receive sms and email reminders when surveys are due.

At baseline, clinician study participants will supervise DNA sample collection and will be prompted to complete a brief survey containing questions about the patient's psychiatric history and severity of illness, current treatment regimen and the treatment intentions of the clinician prior to receiving genetic results. After receiving the results of the Assay, clinician study participants will again be prompted to complete an online study survey containing questions related to the impact of the Genecept Assay on treatment and diagnosis decisions. The subject will continue with treatment as determined by the clinician study participant. At 3 months from baseline, clinician study participants will again be asked to complete an online survey with additional questions related to subsequent changes to the patient's treatment regimen and illness severity since receiving/implementing the results of the Assay.

The subject will also be prompted to complete surveys at baseline, 1 month from the receipt of the genetic results and 3 months from the receipt of the genetic results. These surveys include questions about the patient's psychiatric symptoms, quality of life and medication side effects. The 3 month patient assessment will also include a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Clinician Study Participants:

* Valid National Provider Identifier (NPI) number and prescribing privileges
* Signed electronic informed consent
* Signed requisitions form for order of Genecept Assay
* Requisition form includes indication of diagnosis of depression or anxiety for patient

Subject Study Participants:

* Ability to complete electronic informed consent; includes:

  * access to appropriate technology (i.e. internet-connected device, internet connection),
  * cognitively competent
* > or = 18 years old at time of DNA sample collection
* Indication of diagnosis of depression or anxiety on requisition form

Exclusion Criteria:

Clinician Study Participants:

* Inability to complete online questionnaires

Subject Study Participants:

* Inability to complete online questionnaires;includes:

  * lack of access to appropriate technology (i.e. internet-connected device, internet connection),
  * cognitive impairment
* < 18 years old at time of DNA sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herb Harris, MD, PhD, Principal Investigator — Genomind, LLC
Locations (1):
- Genomind, LLC, Chalfont, Pennsylvania, United States

REFERENCES:
- [Derived] Brennan FX, Gardner KR, Lombard J, Perlis RH, Fava M, Harris HW, Scott R. A Naturalistic Study of the Effectiveness of Pharmacogenetic Testing to Guide Treatment in Psychiatric Patients With Mood and Anxiety Disorders. Prim Care Companion CNS Disord. 2015 Apr 16;17(2):10.4088/PCC.14m01717. doi: 10.4088/PCC.14m01717. eCollection 2015. PMID 26445691

RESULTS

PARTICIPANT FLOW:
Groups:
- Clincian-Reported Outcomes: Prescribing clinicians responsible for the treatment of patients age 18 and older with a primary diagnosis of Major Depressive Disorder or Generalized Anxiety disorder, and for whom the Genecept Assay has been utilized to perform genetic testing.
  Genecept Assay: Genetic test which analyzes seven pharmacodynamic and three pharmacokinetic genes important in psychiatric disorders
- Patient-Reported Measures: Patients age 18 and older with a diagnosis of Major Depressive Disorder or Generalized Anxiety disorder who receive genetic testing using the Genecept Assay and used self-reported patient scales to measure clinical improvements.
Period: Overall Study
Arm/Group | Clincian-Reported Outcomes | Patient-Reported Measures
Started | 625 | 60
Completed | 625 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clinician-Reported Outcomes
Number analyzed (Participants) | 625
Age, Continuous [Mean (Full Range); unit: years] | 40.5 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants] — Clinicians completed assessments for 625 patients. In addition, 197 patients completed self-assessments; however, 137 of these assessments corresponded with the clinicians'. The remaining 60 assessments that differed from the clinicians' were included in the data (n=625+60=685). Baseline measures only came from clinician assessments, explaining n=625.
  Participants
    Female | 412
    Male | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Baseline measures only came from clinician assessments, explaining n=625.
  Participants
    Hispanic or Latino | 25
    Not Hispanic or Latino | 600
    Unknown or Not Reported | 0
Current Smoker [Number; unit: participants] — Baseline measures only came from clinician assessments, explaining n=625.
  participants
    Current Smoker | 36
    Not a smoker | 227
    Unknown | 362
Marital Status [Number; unit: participants] — Baseline measures only came from clinician assessments, explaining n=625.
  participants
    Married | 177
    Divorced/Separated | 53
    Single | 118
    Widowed | 1
    Unknown | 276
Education [Number; unit: participants] — Baseline measures only came from clinician assessments, explaining n=625.
  participants
    >College degree | 145
    Some college | 140
    High school diploma | 50
    No high school diploma | 6
    Unknown | 284
Employment Status [Number; unit: participants] — Baseline measures only came from clinician assessments, explaining n=625.
  participants
    Full-time | 182
    Part-time | 39
    Unemployed/disabled/leave of absence | 83
    Student | 33
    Retired | 12
    Unknown | 276
Annual Income [Number; unit: participants] — Baseline measures only came from clinician assessments, explaining n=625.
  participants
    > $75,000 | 62
    $25,000-75,000 | 152
    < $25,000 | 135
    Unknown | 276

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Global Impressions Improvement (CGI-I) Scale at 3 Months
Description: To determine the efficacy of assay-guided treatment (AGT) in terms of illness severity, as measured by change from baseline using the clinician-administered CGI-I scale, which ranges from scores 1-7 (1=very much improved, 7=very much worse since initiation of treatment).
Time Frame: 3 months
Measure: Number; unit: Participants
Groups:
- Clinician's Utilizing Assay Guided Treatment in Psychiatry: Prescribing clinicians responsible for the treatment of patients age 18 and older with a primary diagnosis of Major Depressive Disorder or Generalized Anxiety disorder, and for whom the Genecept Assay has been utilized to perform genetic testing.
  Genecept Assay: Genetic test which analyzes seven pharmacodynamic and three pharmacokinetic genes important in psychiatric disorders
Arm/Group | Clinician's Utilizing Assay Guided Treatment in Psychiatry
Number analyzed (Participants) | 625
Participants
  CGI-I Score 1, 2, or 3 | 545
  CGI-I Score 1 or 2 | 386

2. Secondary Outcome: Efficacy Measured by QIDS-SR16, Q-LES-Q-SF, UKU Side Effects; and SAS at 3 Months
Description: To determine the efficacy of assay-guided treatment (AGT) in terms of illness severity as measured by change from baseline in self-reported patients scales:
  1. Quick Inventory of Depressive Symptoms (QIDS-SR16) scale; scores range from 0-27, 0 means no depression and 27 means very severe depression
  2. Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) scale; scores range from 0-100 and greater scores correspond with greater satisfaction with quality of life
  3. Undersøgelser (UKU) scale that measures degree of side effects from total scores ranging from 0-100; 0-40 refers to low side effects and 81-100 referring to high side effects rating
  4. the Zung Self-Rated Anxiety (SAS) scale measures anxiety severity using the total scores ranging from 20-80; 20-44 being normal and 75-80 meaning most severe
Time Frame: 3 months
Population: Only 197 patients completed self-assessments at 3 months.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Clinician's Utilizing Assay Guided Treatment in Psychiatry
Number analyzed (Participants) | 197
Scores on a scale
  QIDS-SR16 | 7.8 (0.75)
  Q-LES-Q-SF | 50.0 (1)
  UKU: Side Effects | 19.2 (2)
  SAS | 35.9 (0.5)

ADVERSE EVENTS:
Groups:
- Patient-Reported Outcomes: Patients age 18 and older with a diagnosis of Major Depressive Disorder or Generalized Anxiety disorder who receive genetic testing using the Genecept Assay and used self-reported patient scales to measure clinical improvements.
Arm/Group | Clinician-Reported Outcomes | Patient-Reported Outcomes
Serious Adverse Events (participants affected / at risk) | 0/625 | 0/60
Other Adverse Events (participants affected / at risk) | 0/625 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes